CLINICAL TRIAL: NCT06115993
Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Single Ascending Doses and Multiple Doses of AHB-137 in Healthy Participants and HBeAg-negative CHB Patients Receiving Stable Nucleos(t)Ide Analogues (NAs) Treatment
Brief Title: A Study to Evaluate the Safety and Efficacy of AHB-137 in Healthy Participants and HBeAg-negative Chronic Hepatitis B (CHB) Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ausper Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB-10-8002
Record Dates: First submitted 2023-10-11; First posted 2023-11-03 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part Ia: dosing in healthy participants (Experimental): SAD of 75 mg, 150 mg, 300 mg and 450 mg AHB-137 and MAD of 150 mg and 300 mg AHB-137 by subcutaneous injections within a month in healthy participants.
  Interventions: Drug: AHB-137 injection; Drug: Placebo
- Part Ib: dosing in CHB participants (Experimental): Dose escalation cohort: MAD of 150 mg and 300 mg AHB-137 by subcutaneous injections within a month in CHB participants who are under stable NAs therapy.
  Dose expansion cohort: Multiple doses of 300 mg AHB-137 by subcutaneous injections within a month in CHB participants who are under stable NAs therapy.
  Interventions: Drug: AHB-137 injection; Drug: Placebo
- Part IIa: proof of concept (Experimental): Multiple doses of 225 mg or 300 mg AHB-137 by subcutaneous injections within 24 weeks in CHB participants who are under stable NAs therapy.
  Interventions: Drug: AHB-137 injection

INTERVENTIONS:
Drug: AHB-137 injection — AHB-137 injection will be administered subcutaneously.
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Part Ia: dosing in healthy participants; Part Ib: dosing in CHB participants

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of AHB-137 subcutaneous injection in healthy participants after single and multiple doses, and evaluate the preliminary efficacy of AHB-137 in CHB participants after up to 24 weeks of treatment as a proof-of-concept.

DETAILED DESCRIPTION:
This study is a three-part study of AHB-137, including Part Ia, Part Ib and Part IIa. Part Ia evaluates the safety, tolerability, pharmacokinetics of AHB-137 following single-ascending doses (SAD) and multiple-ascending doses (MAD) in healthy participants. Part Ib is a multiple-dose study to assess the safety, tolerability, pharmacokinetics, and initial efficacy of AHB-137 in CHB participants following weekly dosing for 4 weeks with two loading doses in the first two weeks. Part IIa is a multiple-dose study to evaluate the preliminary efficacy, safety and pharmacokinetics of AHB-137 in CHB participants following weekly dosing for 24 weeks with two loading doses in the first two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants are required to meet all the following inclusion criteria in order to be enrolled in the study (Part Ia):

  1. The participants voluntarily participate in the study, and sign the Informed Consent Form (ICF) prior to screening;
  2. The participants are able to comply with all the protocol requirements;
  3. The participants (and partners) are willing to take effective contraceptive measures from the screening until at least 6 months after the last dosing;
  4. Male or female aged 18-55 when signing ICF;
  5. Body Mass Index (BMI) between 18 to 28 kg/m2 (inclusive) and body weight equal to or over 50 kg for male and 45 kg for female;
  6. Vital signs and physical examination are normal, or abnormal values are not clinically significant.
* CHB participants are required to meet all the following inclusion criteria in order to be enrolled in the study (Part Ib and part IIa):

  1. The participants voluntarily participate in the study, and sign the Informed Consent Form (ICF) prior to screening;
  2. The participants are able to comply with all the protocol requirements;
  3. The participants (and partners) are willing to take effective contraceptive measures from the screening until at least 6 months after the last dosing;
  4. Male or female aged 18-65 when signing ICF;
  5. Body Mass Index (BMI) between 18 to 32 kg/m2 (inclusive) and body weight equal to or over 45 kg for male and 40 kg for female;
  6. participants who have documented chronic HBV infection equal to or above 6 months prior to screening.
  7. Stable treatment of HBeAg negative CHB participants;
  8. Currently receiving single-agent treatment with stable NAs (TDF, TAF, or ETV) for at least 6 months and no changes in the NAs treatment regimen are planned during the trial;
  9. Serum ALT≤2×ULN, HBV DNA < 100 IU/mL. Dose increasing stage of Ib: 100 IU/mL <HBsAg≤1000 IU/mL; Dose expansion stage of Ib: 1000 IU/ml < HBsAg≤3000 IU/mL at screening; IIa phase: 100 IU/ml < HBsAg≤ 3000 IU/mL at screening;
  10. Participants who are willing and able to terminate NA treatment according to the protocol in IIa stage.

Exclusion Criteria:

* Healthy participants are required to not meet any of the exclusion criteria in order to be enrolled in the study (Part Ia):

  1. Any suspicat screening ion of drug component allergy, or allergic constitution (various drug and food allergy, and judged by the investigator to be clinically significant) in participants;
  2. Blood donation or blood loss not less than 400 mL within 12 weeks before screening;
  3. Drug administration that change the activity of liver enzymes within 28 days prior to screening;
  4. Receipt of another investigational drug or device within 3 months before first dosing (interventional treatment);
  5. Clinically significant electrocardiogram (ECG) abnormalities on screening ECG;
  6. TdP high-risk factors (hypokalemia, hypomagnesemia, decompensated heart failure and acute myocardial infarction), and QTc interval above 450 msec in participants (judged by investigator based on actual screening conditions);
  7. Pregnant (positive pregnancy test), recently ready to conceive, or lactating female;
  8. Clinically significant lab examination abnormalities, or other clinically significant diseases discovered within 12 months before screening, including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrinological, tumor, pulmonary, immune, mental, or cardiovascular and cerebrovascular diseases;
  9. Any acute disease or concomitant medication occurred during screening to the first dosing;
  10. Alcohol consumption, or positive alcohol test 24 hours before drug dosing;
  11. Positive test for urinalysis (including Morphine, Cannabis) in participants;
  12. Other factors resulting in participant becoming unsuitable for the study, determined by the investigator.
* CHB participants are required to not meet any of the exclusion criteria in order to be enrolled in the study (Part Ib and Part IIa):

  1. Any suspicion of drug component allergy, or allergic constitution (various drug and food allergy, and judged by the investigator to be clinically significant) in participants;
  2. Blood donation or blood loss more than 400 mL within 12 weeks before screening; Blood transfusion; Blood donation or blood loss not less than 200 mL within 1 month before screening;
  3. Any oligonucleotide or siRNA treatments within 12 months before first dosing;
  4. Any immunosuppressing, immunomodulator (e.g. Thymosin) or cytotoxic drug administrations within 6 months before first dosing; Vaccination within 1 month in prior of screening, or plan to take any vaccines during the study;
  5. Receiving anticoagulant therapy for Ib phase (e.g., Warfarin, Factor Xa Inhibitors or antiplatelet drugs such as Clopidogrel);
  6. Any clinically significant liver diseases, including but not limited to hepatitis caused by other pathogenic infections, hemochromatosis, Wilson disease, primary biliary cirrhosis, autoimmune liver diseases, alcoholic liver disease, severe non-alcoholic fatty liver disease, Drug-induced liver injury, etc.;
  7. Personal history of cirrhosis or progressive hepatic fibrosis (e.g., the participant undergoes hepatic histopathological examination, which indicates cirrhosis, or undergoes endoscopic examination indicating esophagogastric varices);
  8. Confirmation or suspicion of decompensated hepatitis B cirrhosis, including but not limited to hepatic encephalopathy, hepatorenal syndrome, esophageal and gastric variceal bleeding, ascites, primary hepatocellular carcinoma, etc.;
  9. History of malignancy within the past 5 years, except for certain tumors that can be cured by surgical resection (e.g., non-melanoma skin cancer, cervical intraepithelial neoplasia, thyroid neoplasm, breast tumor, etc. that have been treated without signs of recurrence);
  10. Combined sever diseases of circulation, digestion, respiration, urinary, blood, metabolism, immune, nervous system, etc.;
  11. Participants for IIa phase with high-risk factors for TdP (hypokalemia, hypomagnesemia, decompensated heart failure, and acute myocardial infarction), baseline QTc interval longer than 450 ms (determined by the researchers based on actual screening);
  12. Acute infection within 2 weeks prior to screening;
  13. Receipt of another investigational drug or device within 1 month before screening (interventional treatment);
  14. Laboratorial examination: blood platelet counts<90 x 10^9/L, absolute neutrophil count<1.3 x 10^9/L, hemoglobin<90 g/L, serum total bilirubin ≥2 x ULN, albumin<30 g/L, creatinine clearance rate (calculated by MDRD formula) ≤60 mL/min, PT/INR>1.5;
  15. Alpha-fetoprotein (AFP) >70 ug/L, or imaging suspicion of malignant hepatic space-occupying;
  16. HCV antibody/HCcAg positive, AIDS antigen/antibody positive, or Treponema Pallidum antibody positive and Rapid Plasma Reagin (RPR) or Toluidine Red Unheated Serum Test (TRUST) positive, or Hepatitis D antibody positive;
  17. LSM≥12.4 kPa when screening;
  18. Pregnant (positive pregnancy test) or lactating female;
  19. Positive test for urinalysis (including Morphine, Cannabis) or alcohol test in participants;
  20. Other factors results in unsuitable for the study, determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of healthy participants with TEAEs, SAEs | Up to 30 days for SAD; up to 113 days for MAD
Number of healthy participants with clinically significant changes in laboratory parameters | Up to 30 days for SAD; up to 113 days for MAD
Number of healthy participants with clinically significant changes in vital signs | Up to 30 days for SAD; up to 113 days for MAD
Number of healthy participants with clinically significant changes in ECG | Up to 30 days for SAD; up to 113 days for MAD
Number of healthy participants with ADA | Up to 30 days for SAD; up to 113 days for MAD
The pharmacokinetic profile of AHB-137 in healthy participants: the Cmax of AHB-137 | Up to 30 days for SAD; up to 113 days for MAD
The pharmacokinetic profile of AHB-137 in healthy participants: Tmax of AHB-137 | Up to 30 days for SAD; up to 113 days for MAD
The pharmacokinetic profile of AHB-137 in healthy participants: AUC of AHB-137 | Up to 30 days for SAD; up to 113 days for MAD
The pharmacokinetic profile of AHB-137 in healthy participants: t1/2 of AHB-137 | Up to 30 days for SAD; up to 113 days for MAD
Number of CHB participants with TEAEs, SAEs | Up to 113 days for Ib
Number of CHB participants with clinically significant changes in laboratory parameters | Up to 113 days for Ib
Number of CHB participants with clinically significant changes in vital signs | Up to 113 days for Ib
Number of CHB participants with clinically significant changes in ECG | Up to 113 days for Ib
Proportion of participants achieving HBsAg lower than LLOQ (0.05 IU/mL) and HBV DNA lower than LLOQ at the end of treatment with AHB-137, regardless of whether HBsAg seroconversion is observed | At week 24 for IIa

SECONDARY OUTCOMES:
The anti-HBV efficacy of AHB-137 in CHB participants: evaluate the serum levels of HBV DNA, HBsAg, HBV RNA, HBsAb, HBeAb | Up to 113 days for Ib; Up to 72 weeks for IIa
Evaluate the serum levels of sensitive HBsAg (LLOQ ≤0.005 IU/mL) and HBcrAg. | Up to 72 weeks for IIa
The pharmacokinetic profile of AHB-137 in CHB participants: the Cmax of AHB-137 | up to 113 days for Ib; Up to 48 weeks for IIa
The pharmacokinetic profile of AHB-137 in CHB participants: Tmax of AHB-137 | up to 113 days for Ib; Up to 48 weeks for IIa
The pharmacokinetic profile of AHB-137 in CHB participants: AUC of AHB-137 | up to 113 days for Ib; Up to 48 weeks for IIa
The pharmacokinetic profile of AHB-137 in CHB participants: t1/2 of AHB-137 | up to 113 days for Ib; Up to 48 weeks for IIa
Number of CHB participants with ADA | Up to113 days for Ib; Up to 48 weeks for IIa
Number of CHB participants with TEAEs, SAEs | Up to 72 weeks for IIa
Number of CHB participants with clinically significant changes in laboratory parameters, ECG, and vital signs | Up to 72 weeks for IIa
Proportion of CHB participants achieving HBsAg lower than LLOQ and HBV DNA lower than LLOQ during or after 24-week treatment, regardless of whether HBsAg seroconversion is observed | Up to 72 weeks for IIa
Proportion of CHB participants meeting the discontinuation criteria for NA treatment | At 48 weeks for IIa
Sequencing of the Viral DNA and/or viral RNA analysis for detection of drug resistance in the target region of AHB-137 | Up to 113 days for Ib; Up to 72 weeks for IIa

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Principal Investigator — The First Hospital of Jilin University; Junqi Niu, Principal Investigator — The First Hospital of Jilin University
Locations (3):
- China (3):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - The First Hospital of Jilin University, Jilin

IPD SHARING:
Plan to Share IPD: No